CLINICAL TRIAL: NCT03125382
Title: PORTuguese Research on Telemonitoring With CareLink® (PORTLink)
Acronym: PORTLink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PORTLink
Record Dates: First submitted 2016-05-25; First posted 2017-04-24 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2023-05

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- In office standard visit-New (Active Comparator): Patients with new implants who do not perform device data transmission through Carelink system
  Interventions: Device: In office standard visit
- In office standard visit-Previous (Active Comparator): Patients with previous implants who do not perform device data transmission through Carelink system
  Interventions: Device: In office standard visit
- Carelink - New Implants (Experimental): Patients with new implants who perform device data transmission through Carelink system
  Interventions: Device: Carelink System
- Carelink - Previous Implants (Experimental): Patients with previous implants who perform device data transmission through Carelink system
  Interventions: Device: Carelink System

INTERVENTIONS:
Device: Carelink System — Patients start to perform device data transmission through Carelink system
  Arms: Carelink - New Implants; Carelink - Previous Implants
Device: In office standard visit — Patients start or maintain in office standard visits
  Arms: In office standard visit-New; In office standard visit-Previous

SUMMARY:
Compare use of Carelink system - monitoring system - with traditional in-clinic follow up, in patients with implantable cardiac defibrillator (ICD)

DETAILED DESCRIPTION:
The objective of the PORTLink (PORTuguese Research on Telemonitoring with CareLink), a multicenter randomized study, is to assess the safety, functioning and costs of remote ICD monitoring when compared to traditional in-clinic follow-up. It will evaluate aspects such as the clinician and patient acceptance and satisfaction with the reviewing device data via the website, the complexity for troubleshooting calls to the support center, the utilization of emergency resources by symptomatic patients, the percentage of the unscheduled appointments after a remote interrogation, the levels of anxiety, depression and quality of life, and the main consumed resources with CareLink System.

ELIGIBILITY:
Inclusion Criteria:

* Subject has implanted Medtronic Implantable Cardioverter Defibrillator: CRT-D (Cardiac Resynchronization Therapy - Defibrillator), ICD
* Subject or the subject's caregiver is willing and able to use the Medtronic CareLink Monitor and perform the required duties at home or have a family member or assistant to perform those studies
* Subject has signed a Patient Informed Consent Form from this study

Exclusion Criteria:

* Subject has medical condition(s) that would limit study participation (e.g. hearing or speech impaired with no family member or assistant available)
* Subject is less than 18 years of age
* Subject is enrolled or intends to participate in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mário Oliveira, Doctor, Principal Investigator — Centro Hospitalar Lisboa Central
Locations (6):
- Portugal (6):
  - Hospital Hospitalar do Algarve, Faro
  - Centro Hospitalar de Alto Ave - Unidade de Guimarães, Guimarães
  - Centro Hospitalar Lisboa Central- Hospital de Santa Marta, Lisbon
  - Centro Hospitalar do Porto, Porto
  - Centro Hospitalar de Setúbal, Setúbal
  - Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start - 01 Apr 2012 Recruitment end - 30 Apr 2015
  Location - In Hospital
Pre-assignment Details: There were 7 screening failures;
Period: Randomization
Arm/Group | In Office Standard Visit-New | In Office Standard Visit-Previous | Carelink - New Implants | Carelink - Previous Implants
Started (Randomization) | 38 | 32 | 37 | 34
Completed | 37 | 28 | 35 | 34
Not Completed | 1 | 4 | 2 | 0
Not completed — screening failure | 1 | 4 | 2 | 0
Period: Follow-up
Arm/Group | In Office Standard Visit-New | In Office Standard Visit-Previous | Carelink - New Implants | Carelink - Previous Implants
Started | 37 | 28 | 35 | 34
Completed | 35 | 22 | 31 | 31
Not Completed | 2 | 6 | 4 | 3
Not completed — Death | 1 | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 4 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In Office Standard Visit-New | In Office Standard Visit-Previous | Carelink - New Implants | Carelink - Previous Implants | Total
Number analyzed (Participants) | 37 | 28 | 35 | 34 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.3) | 62.0 (15.2) | 56.5 (13.7) | 63.8 (10.9) | 59.9 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 10 | 4 | 27
  Male | 30 | 22 | 25 | 30 | 107
Type of Device [Count of Participants; unit: Participants]
  Implantable Cardioverter Defibrillator | 26 | 19 | 27 | 24 | 96
  Cardiac Resynchronization Therapy Defibrillator | 11 | 9 | 8 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient Satisfied or Very Satisfied With Carelink
Description: through the semi-quantitative evaluation of patient satisfaction with Carelink System and their preference when compared to traditional in-clinic follow-up, the options were: 1) Very Satisfied; 2) Satisfied; 3) Not Satisfied nether Unsatisfied; 4) Unsatisfied; 5)Very Unsatisfied
Time Frame: 12 months visit
Population: Only applicable for Carelink arms
Measure: Count of Participants; unit: Participants
Arm/Group | Carelink - New Implants | Carelink - Previous Implants
Number analyzed (Participants) | 35 | 34
Participants | 34 | 34

2. Secondary Outcome: Number of Device Related Adverse Events
Description: compare number of Device-related Adverse Events
Time Frame: 12 months visit
Measure: Count of Participants; unit: Participants
Arm/Group | In Office Standard Visit-New | In Office Standard Visit-Previous | Carelink - New Implants | Carelink - Previous Implants
Number analyzed (Participants) | 37 | 28 | 35 | 34
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Physician Satisfaction With Carelink: Total Number of Transmissions With Satisfaction Ratings
Description: Through the semi-quantitative evaluation of physician satisfaction with CareLink System.
  Used rating: "Very Satisfied"; "Satisfied"; "neither satisfied nor dissatisfied"; "dissatisfied" and "very dissatisfied"
Time Frame: 12 months visit
Measure: Number; unit: satisfaction at each transmission
Arm/Group | Carelink - New Implants | Carelink - Previous Implants
Number analyzed (Participants) | 35 | 34
satisfaction at each transmission
  very satisfied | 98 | 80
  satisfied | 25 | 47
  neither satisfied nor dissatisfied | 0 | 0
  dissatisfied | 0 | 0
  Neither satisfied nor dissatisfied | 0 | 0

4. Secondary Outcome: Health Care Consumed Resources Between Groups Relative to Unscheduled Visits
Description: Number of in office unscheduled visits will be calculated per arm and compared with each other
Time Frame: 12 months visit
Population: It was pre-specified to combine "In Office Standard Visit-New" and "In Office Standard Visit-Previous" Arms/Groups and "Carelink - New Implants" and "Carelink - Previous Implants" Arms/Groups for this analysis
Measure: Mean (Standard Deviation); unit: visits
Groups:
- In Office Standard Visit: Patients with new implants who do not perform device data transmission through Carelink system
  In office standard visit: Patients start or maintain in office standard visits
- Carelink: Patients with new implants who perform device data transmission through Carelink system
  Carelink System: Patients start to perform device data transmission through Carelink system
Arm/Group | In Office Standard Visit | Carelink
Number analyzed (Participants) | 65 | 69
visits | 1.1 (0.9) | 0.4 (0.6)

5. Secondary Outcome: Compare Patient Consumed Resources Between Groups
Description: Attribute patient travel costs to low, middle and high costs and then compare patient travel costs between the group with in office visits versus Carelink, measured at baseline
Time Frame: Baseline
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- In Office Standard Visit: Patients with previous or new implants who do not perform device data transmission through Carelink system
  In office standard visit: Patients start or maintain in office standard visits
- Carelink: Patients with previous or new implants who perform device data transmission through Carelink system
  Carelink System: Patients start to perform device data transmission through Carelink system
Arm/Group | In Office Standard Visit | Carelink
Number analyzed (Participants) | 64 | 69
Participants
  Up to 5 € | 23 | 23
  5 - 15 € | 21 | 26
  More than 15€ | 20 | 20

6. Secondary Outcome: Compare Patient Consumed Resources Between Groups
Description: Patient time consumption in visits between the groups at baseline visit
  Arms were combine:
  * In office standard visit combined: Office Standard Visit-New + In Office Standard Visit-Previous
  * Carelink combine: Carelink - New Implants & Carelink - Previous
Time Frame: Baseline
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | In Office Standard Visit | Carelink
Number analyzed (Participants) | 65 | 69
Minutes
  Travel time | 30 [15 to 60] | 30 [20 to 60]
  Time at the hospital | 80 [50 to 110] | 95 [60 to 140]

7. Secondary Outcome: Improvement in Quality of Life
Description: Health-related quality of life was measured with an adapted version of the SF-12 questionnaire, a 12-item generic measure derived from the Short-Form 36. It evaluates physical functioning, limitations due to physical health problems, bodily pain, energy/fatigue, social functioning, limitations due to emotional problems, and psychological distress and well-being. Physica lcomponent summary and mental component summary measures were estimated, with higher scores indicating better health status (range from 0 to 100).
  Mental health wellbeing was measured with the Hospital Anxiety and Depression Scale (HADS), which consists of a series of 14 questions, seven related to anxiety (HAD-A) plus other seven questions related to depression (HAD-D). Scores of 0-7 for the two subscales are regarded as normal, scores of 8-10 suggest the presence of a mood disorder and scores ≥11 suggest a probable mood disorder.
Time Frame: 12 months visit
Population: It was pre-specified to combine "In Office Standard Visit-New" and "In Office Standard Visit-Previous" Arms/Groups and "Carelink - New Implants" and "Carelink - Previous Implants" Arms/Groups for this analysis
  Within each group, nonparametric Wilcoxon rank-sum test for paired samples was used to determine the statistical significance of changes on anxiety, depression and SF-12 scores. Changes in HADS anxiety and depression scores, SF-12 were evaluated by analysis of covariance (ANCOVA) models
Measure: Mean (95% Confidence Interval); unit: score change
Arm/Group | In Office Standard Visit | Carelink
Number analyzed (Participants) | 65 | 69
score change
  HADS anxiety | 0 [-3 to -0] | 0 [-3 to 1]
  HADS depression | 0 [-2 to 1] | 0 [-2 to 1]
  SF12 physical component | -1.1 [-8.1 to 2.6] | 0.0 [-4.5 to 4.9]
  SF12 mental component | 0.4 [-3.9 to 7.5] | 0.0 [-9.5 to 5.6]

8. Secondary Outcome: Number of Unanticipated Serious Adverse Device Effects (USADE) Rate
Description: compare number of Unanticipated Serious Adverse Device Effects (USADE)
  Arms were combine:
  * In office standard visit combined: Office Standard Visit-New + In Office Standard Visit-Previous
  * Carelink combine: Carelink - New Implants & Carelink - Previous
Time Frame: 12 months visit
Population: as for outcome 4
Measure: Number; unit: adverse event
Arm/Group | In Office Standard Visit | Carelink
Number analyzed (Participants) | 65 | 69
adverse event | 6 | 4

ADVERSE EVENTS:
Time Frame: 12 months visit
Groups:
- In Office Standard Visit-New: Patients with new implants who do not perform device data transmission through Carelink system
  In office standard visit: Patients start or maintain office standard visits
Arm/Group | In Office Standard Visit-New | In Office Standard Visit-Previous | Carelink - New Implants | Carelink - Previous Implants
All-Cause Mortality (participants affected / at risk) | 1/37 | 2/28 | 1/35 | 2/34
Serious Adverse Events (participants affected / at risk) | 1/37 | 2/28 | 1/35 | 2/34
Other Adverse Events (participants affected / at risk) | 1/37 | 2/28 | 0/35 | 1/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Office Standard Visit-New (N=37) | In Office Standard Visit-Previous (N=28) | Carelink - New Implants (N=35) | Carelink - Previous Implants (N=34)
Death (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — unknown death cause
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — resulted in the death
Exarcebation chronic kidney disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — resulted in the death
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — resulted in the death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In Office Standard Visit-New (N=37) | In Office Standard Visit-Previous (N=28) | Carelink - New Implants (N=35) | Carelink - Previous Implants (N=34)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
AF with fast ventricular response (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decompesated cardiac failure episode (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No